CLINICAL TRIAL: NCT04702568
Title: A Phase 2, Open-Label Study to Evaluate the Long-term Safety of Oral BCX9930 in Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: A Long-Term Safety Study of BCX9930 in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCX9930-201; 2020-000501-93 (EudraCT Number)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; PNH
Keywords: BCX9930; Factor D inhibitor; PNH; paroxysmal Nocturnal Hemoglobinuria; oral treatment
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab; ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Complement Component 5 (C5) Inhibitor (C5-INH) Naïve Group (Experimental): This group included participants who, prior to enrolling in their previous BCX9930 study, were either naïve to eculizumab or ravulizumab treatment, or naive to treatment with any complement inhibitor therapy (or had received no treatment in the prior 12 months), and with anemia due to ongoing intravascular hemolysis.
  Interventions: Drug: BCX9930
- C5 INH Inadequate Response Group (Experimental): This group included participants who, prior to enrolling in their previous BCX9930 study, were receiving stable treatment with eculizumab or ravulizumab and had an inadequate response to that therapy (ie, residual anemia and/or ongoing need for transfusion). Depending on the prior study, participants may have continued the C5 inhibitor, with BCX9930 provided as an add-on therapy.
  Interventions: Drug: BCX9930; Drug: Eculizumab; Drug: Ravulizumab

INTERVENTIONS:
Drug: BCX9930 — BCX9930 for oral administration
Drug: Eculizumab — Administered at stable dose at the time of study entry
  Arms: C5 INH Inadequate Response Group
Drug: Ravulizumab — Administered at stable dose at the time of study entry
  Arms: C5 INH Inadequate Response Group

SUMMARY:
This study was designed to evaluate the long-term safety of daily oral treatment with BCX9930 in participants who had participated in a previous BCX9930 trial for PNH and showed a benefit of treatment as determined by the Investigator. The study allowed continued access to BCX9930 for enrolled participants. The study also evaluated the long-term effectiveness and impact on quality of life and general well-being of BCX9930 treatment, and the participant's satisfaction with the medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female participants
* Successfully participated in a previous BCX9930 study of PNH and experienced improvement in their PNH

Exclusion Criteria:

* Apart from a diagnosis of PNH, any clinically significant medical or psychiatric condition or medical history, other than those associated with PNH disease, that, in the opinion of the Investigator or Sponsor, would interfere with the participant's ability to participate in the study or participation would increase the risk for that participant
* Pregnant, planning to become pregnant, or having been pregnant within 90 days of Day 1, or lactating

Note: Other protocol-defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morag Griffin, MBChB, Principal Investigator — Leeds Teaching Hospitals NHS Trust, Leeds, UK
Locations (5):
- Study Center, Vienna, Austria
- South Africa (3):
  - Study Center, Bloemfontein
  - Study Center, Cape Town
  - Study Center, Pretoria
- Study Center, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had participated in previous BCX9930 trials (BCX9930-101 [NCT04330534], BCX9930-202 [NCT05116774], or BCX9930-203 [NCT05116787]) for Paroxysmal Nocturnal Hemoglobinuria (PNH) and showed a benefit of treatment as determined by the investigator were enrolled in this long-term safety trial.
Groups:
- Complement Component 5 (C5) Inhibitor (C5-INH) Naïve Group: This group included participants who, prior to enrolling in their previous BCX9930 study, were either naïve to eculizumab or ravulizumab treatment, or naive to treatment with any complement inhibitor therapy (or had received no treatment in the prior 12 months), and with anemia due to ongoing intravascular hemolysis. Participants were to commence treatment at the same BCX9930 dose level and regimen last administered to that individual in the prior study. Per last protocol amendment, all participants received BCX9930 400 milligrams (mg) orally twice daily (BID). Treatment duration was up to 144 weeks.
- C5-INH Inadequate Response Group: This group included participants who, prior to enrolling in their previous BCX9930 study, were receiving stable treatment with eculizumab or ravulizumab and had an inadequate response to that therapy (ie, residual anemia and/or ongoing need for transfusion). Depending on the prior study, participants may have continued the C5 inhibitor, with BCX9930 provided as an add-on therapy. Participants were to commence treatment at the same BCX9930 dose level and regimen last administered to that individual in the prior study. Per last protocol amendment, all participants received BCX9930 400 mg orally BID. Treatment duration was up to 144 weeks.
Period: Overall Study
Arm/Group | Complement Component 5 (C5) Inhibitor (C5-INH) Naïve Group | C5-INH Inadequate Response Group
Started | 12 | 7
Completed | 0 | 0
Not Completed | 12 | 7
Not completed — Transitioned to the BCX9930-205 roll-over study | 10 | 4
Not completed — Pregnancy | 1 | 0
Not completed — Bone marrow transplant | 1 | 0
Not completed — Withdrawn due to Investigator decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 capsule or tablet of study drug.
Groups:
- C5-INH Naïve Group: This group included participants who, prior to enrolling in their previous BCX9930 study, were either naïve to eculizumab or ravulizumab treatment, or naive to treatment with any complement inhibitor therapy (or had received no treatment in the prior 12 months), and with anemia due to ongoing intravascular hemolysis. Participants were to commence treatment at the same BCX9930 dose level and regimen last administered to that individual in the prior study. Per last protocol amendment, all participants received BCX9930 400 mg orally BID. Treatment duration was up to 144 weeks.
- Total: Total of all reporting groups
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (7.82) | 44.6 (18.59) | 34.9 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 9 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related in a participant or clinical investigation participant who administered a pharmaceutical product regardless of its causal relationship to the study treatment. An AE was considered treatment-emergent if its start date and time was on or after the date and time of first on-study dose of study drug.
Time Frame: From first dose of study drug up to 3 weeks after last dose (Week 147)
Population: The safety population included all participants who received at least 1 capsule or tablet of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants | 12 | 7

2. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Fatigue
Description: Data was reported for number of participants with clinical PNH symptom of fatigue. The severity of clinical PNH symptom of fatigue was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: The mITT (modified intent-to-treat) population included all participants who received at least 1 capsule or tablet of study drug and had post baseline assessment of PNH symptoms and/or laboratory data. Participants with available data at each visit were included.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 8 | 4
  Baseline-mild | 3 | 2
  Baseline-moderate | 0 | 1
  Baseline-severe | 1 | 0
  Week 24-none | 10 | 3
  Week 24-mild | 2 | 3
  Week 24-moderate | 0 | 1
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 6 | 2
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 2 | 0
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 0 | 1
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 0 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 7 | 1
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 1 | 2
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 6 | 2
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 2 | 0
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 1
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 8 | 2
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 0
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 1
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0

3. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Dyspnea
Description: Data was reported for number of participants with clinical PNH symptom of Dyspnea. The severity of clinical PNH symptom of Dyspnea was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 11 | 6
  Baseline-mild | 1 | 1
  Baseline-moderate | 0 | 0
  Baseline-severe | 0 | 0
  Week 24-none | 11 | 7
  Week 24-mild | 1 | 0
  Week 24-moderate | 0 | 0
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 6 | 2
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 2 | 1
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 0 | 0
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 0 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 7 | 2
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 1 | 1
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 7 | 2
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 0 | 0
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 1 | 1
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 0
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 8 | 2
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 1
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0

4. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Chest Pain/Discomfort
Description: Data was reported for number of participants with clinical PNH symptom of Chest pain/discomfort. The severity of clinical PNH symptom of chest pain/discomfort was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 12 | 7
  Baseline-mild | 0 | 0
  Baseline-moderate | 0 | 0
  Baseline-severe | 0 | 0
  Week 24-none | 12 | 7
  Week 24-mild | 0 | 0
  Week 24-moderate | 0 | 0
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 7 | 2
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 1 | 1
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 0 | 0
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 0 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 7 | 2
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 1 | 0
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 1
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 7 | 3
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 1 | 0
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 0
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 8 | 3
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 0
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0

5. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Difficulty Swallowing
Description: Data was reported for number of participants with clinical PNH symptom of difficulty swallowing. The severity of clinical PNH symptom of difficulty swallowing was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 11 | 6
  Baseline-mild | 1 | 1
  Baseline-moderate | 0 | 0
  Baseline-severe | 0 | 0
  Week 24-none | 12 | 7
  Week 24-mild | 0 | 0
  Week 24-moderate | 0 | 0
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 6 | 2
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 2 | 1
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 0 | 0
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 0 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 7 | 2
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 1 | 1
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 7 | 2
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 1 | 1
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 0
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 8 | 3
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 0
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0

6. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Abdominal Pain
Description: Data was reported for number of participants with clinical PNH symptom of abdominal pain. The severity of clinical PNH symptom of abdominal pain was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 10 | 7
  Baseline-mild | 1 | 0
  Baseline-moderate | 1 | 0
  Baseline-severe | 0 | 0
  Week 24-none | 9 | 6
  Week 24-mild | 2 | 0
  Week 24-moderate | 1 | 1
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 6 | 2
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 1 | 1
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 0 | 0
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 1 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 7 | 2
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 1 | 1
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 7 | 2
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 1 | 1
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 0
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 8 | 3
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 0
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0

7. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Headache
Description: Data was reported for number of participants with clinical PNH symptom of headache. The severity of clinical PNH symptom of headache was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 10 | 7
  Baseline-mild | 2 | 0
  Baseline-moderate | 0 | 0
  Baseline-severe | 0 | 0
  Week 24-none | 11 | 6
  Week 24-mild | 1 | 1
  Week 24-moderate | 0 | 0
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 7 | 2
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 0 | 0
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 1 | 1
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 0 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 8 | 3
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 0 | 0
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 7 | 3
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 1 | 0
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 0
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 8 | 2
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 1
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0

8. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Erectile Dysfunction
Description: Data was reported for number of participants with clinical PNH symptom of erectile dysfunction. The severity of clinical PNH symptom of erectile dysfunction was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none: number analyzed (Participants) | 9 | 2
  Baseline-none | 9 | 2
  Baseline-mild: number analyzed (Participants) | 9 | 2
  Baseline-mild | 0 | 0
  Baseline-moderate: number analyzed (Participants) | 9 | 2
  Baseline-moderate | 0 | 0
  Baseline-severe: number analyzed (Participants) | 9 | 2
  Baseline-severe | 0 | 0
  Week 24-none: number analyzed (Participants) | 9 | 2
  Week 24-none | 9 | 2
  Week 24-mild: number analyzed (Participants) | 9 | 2
  Week 24-mild | 0 | 0
  Week 24-moderate: number analyzed (Participants) | 9 | 2
  Week 24-moderate | 0 | 0
  Week 24-severe: number analyzed (Participants) | 9 | 2
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 1
  Week 48-none | 7 | 1
  Week 48-mild: number analyzed (Participants) | 8 | 1
  Week 48-mild | 1 | 0
  Week 48-moderate: number analyzed (Participants) | 8 | 1
  Week 48-moderate | 0 | 0
  Week 48-severe: number analyzed (Participants) | 8 | 1
  Week 48-severe | 0 | 0
  Week 72-none: number analyzed (Participants) | 8 | 1
  Week 72-none | 7 | 1
  Week 72-mild: number analyzed (Participants) | 8 | 1
  Week 72-mild | 1 | 0
  Week 72-moderate: number analyzed (Participants) | 8 | 1
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 1
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 2
  Week 96-none | 7 | 2
  Week 96-mild: number analyzed (Participants) | 8 | 2
  Week 96-mild | 1 | 0
  Week 96-moderate: number analyzed (Participants) | 8 | 2
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 2
  Week 96-severe | 0 | 0
  Week 120-none: number analyzed (Participants) | 8 | 1
  Week 120-none | 7 | 1
  Week 120-mild: number analyzed (Participants) | 8 | 1
  Week 120-mild | 1 | 0
  Week 120-moderate: number analyzed (Participants) | 8 | 1
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 1
  Week 120-severe | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Hemoglobinuria
Description: Data was reported for number of participants with clinical PNH symptom of Hemoglobinuria.The severity of clinical PNH symptom of hemoglobinuria was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 10 | 7
  Baseline-mild | 0 | 0
  Baseline-moderate | 0 | 0
  Baseline-severe | 0 | 0
  Baseline-missing severity | 2 | 0
  Week 24-none | 11 | 5
  Week 24-mild | 0 | 0
  Week 24-moderate | 0 | 0
  Week 24-severe | 0 | 0
  Week 24-missing severity | 1 | 2
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 6 | 3
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 0 | 0
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 1 | 0
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 0 | 0
  Week 48-missing severity: number analyzed (Participants) | 8 | 3
  Week 48-missing severity | 1 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 7 | 2
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 0 | 1
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 72-missing severity: number analyzed (Participants) | 8 | 3
  Week 72-missing severity | 1 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 6 | 3
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 0 | 0
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 0
  Week 96-missing severity: number analyzed (Participants) | 8 | 3
  Week 96-missing severity | 2 | 0
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 7 | 3
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 0
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0
  Week 120-missing severity: number analyzed (Participants) | 8 | 3
  Week 120-missing severity | 1 | 0

10. Secondary Outcome: Number of Participants With Clinical PNH Symptom Based on Severity: Jaundice
Description: Data was reported for number of participants with clinical PNH symptom of jaundice. The severity of clinical PNH symptom of jaundice was graded as none, mild, moderate and severe based solely on investigator's discretion.
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Baseline-none | 11 | 7
  Baseline-mild | 0 | 0
  Baseline-moderate | 0 | 0
  Baseline-severe | 0 | 0
  Baseline-missing severity | 1 | 0
  Week 24-none | 12 | 7
  Week 24-mild | 0 | 0
  Week 24-moderate | 0 | 0
  Week 24-severe | 0 | 0
  Week 48-none: number analyzed (Participants) | 8 | 3
  Week 48-none | 8 | 3
  Week 48-mild: number analyzed (Participants) | 8 | 3
  Week 48-mild | 0 | 0
  Week 48-moderate: number analyzed (Participants) | 8 | 3
  Week 48-moderate | 0 | 0
  Week 48-severe: number analyzed (Participants) | 8 | 3
  Week 48-severe | 0 | 0
  Week 72-none: number analyzed (Participants) | 8 | 3
  Week 72-none | 8 | 3
  Week 72-mild: number analyzed (Participants) | 8 | 3
  Week 72-mild | 0 | 0
  Week 72-moderate: number analyzed (Participants) | 8 | 3
  Week 72-moderate | 0 | 0
  Week 72-severe: number analyzed (Participants) | 8 | 3
  Week 72-severe | 0 | 0
  Week 96-none: number analyzed (Participants) | 8 | 3
  Week 96-none | 8 | 3
  Week 96-mild: number analyzed (Participants) | 8 | 3
  Week 96-mild | 0 | 0
  Week 96-moderate: number analyzed (Participants) | 8 | 3
  Week 96-moderate | 0 | 0
  Week 96-severe: number analyzed (Participants) | 8 | 3
  Week 96-severe | 0 | 0
  Week 120-none: number analyzed (Participants) | 8 | 3
  Week 120-none | 8 | 3
  Week 120-mild: number analyzed (Participants) | 8 | 3
  Week 120-mild | 0 | 0
  Week 120-moderate: number analyzed (Participants) | 8 | 3
  Week 120-moderate | 0 | 0
  Week 120-severe: number analyzed (Participants) | 8 | 3
  Week 120-severe | 0 | 0

11. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH)
Time Frame: Baseline, Weeks, 24, 48, 72, 96, 120, and 144
Population: Participants in the mITT population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 6
Units per liter (U/L)
  Baseline | 475.6 (210.98) | 248.3 (125.71)
  Change at Week 24: number analyzed (Participants) | 11 | 5
  Change at Week 24 | -46.7 (154.55) | 38.6 (45.51)
  Change at Week 48: number analyzed (Participants) | 8 | 2
  Change at Week 48 | -62.5 (80.97) | 38.5 (65.76)
  Change at Week 72: number analyzed (Participants) | 8 | 2
  Change at Week 72 | -6.1 (238.41) | 163.5 (118.09)
  Change at Week 96: number analyzed (Participants) | 8 | 2
  Change at Week 96 | 237.4 (347.65) | -4.0 (134.35)
  Change at Week 120: number analyzed (Participants) | 8 | 2
  Change at Week 120 | 195.4 (355.03) | 31.0 (125.87)
  Change at Week 144: number analyzed (Participants) | 1 | 0
  Change at Week 144 | -59.0 |

12. Secondary Outcome: Change From Baseline in Hemoglobin
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, and 144
Population: Participants in the mITT population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dl)
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
grams per deciliter (g/dl)
  Baseline | 11.88 (1.688) | 11.53 (1.803)
  Change at Week 24: number analyzed (Participants) | 11 | 6
  Change at Week 24 | 0.75 (1.159) | -1.32 (2.578)
  Change at Week 48: number analyzed (Participants) | 8 | 2
  Change at Week 48 | -0.61 (1.974) | -0.95 (2.333)
  Change at Week 72: number analyzed (Participants) | 8 | 3
  Change at Week 72 | -0.64 (2.327) | -0.93 (1.484)
  Change at Week 96: number analyzed (Participants) | 8 | 2
  Change at Week 96 | -0.33 (1.914) | -0.70 (2.687)
  Change at Week 120: number analyzed (Participants) | 8 | 3
  Change at Week 120 | 0.38 (1.555) | -0.47 (2.098)
  Change at Week 144: number analyzed (Participants) | 1 | 0
  Change at Week 144 | -2.70 |

13. Secondary Outcome: Change From Baseline in Haptoglobin
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 5
grams per liter (g/L)
  Baseline | 0.325 (0.2832) | 0.216 (0.1350)
  Change at Week 24: number analyzed (Participants) | 11 | 5
  Change at Week 24 | 0.000 (0.0447) | -0.082 (0.0844)
  Change at Week 48: number analyzed (Participants) | 8 | 0
  Change at Week 48 | 0.213 (0.1126) |
  Change at Week 72: number analyzed (Participants) | 8 | 2
  Change at Week 72 | 0.025 (0.1165) | -0.210 (0.1414)
  Change at Week 96: number analyzed (Participants) | 8 | 2
  Change at Week 96 | -0.013 (0.0354) | 0.195 (0.4313)
  Change at Week 120: number analyzed (Participants) | 8 | 1
  Change at Week 120 | -0.013 (0.0354) | -0.100

14. Secondary Outcome: Change From Baseline in Reticulocytes
Time Frame: Baseline, Weeks 24, 48, 72, 96, and 120
Population: Participants in the mITT population with available data were analyzed
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter (μL)
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
10^6 cells per microliter (μL)
  Baseline | 0.1066 (0.02363) | 0.0889 (0.03939)
  Change at Week 24: number analyzed (Participants) | 11 | 6
  Change at Week 24 | 0.0164 (0.02339) | 0.0913 (0.09144)
  Change at Week 48: number analyzed (Participants) | 8 | 2
  Change at Week 48 | 0.0048 (0.03518) | 0.0507 (0.03161)
  Change at Week 72: number analyzed (Participants) | 8 | 3
  Change at Week 72 | 0.0044 (0.03643) | 0.0463 (0.03008)
  Change at Week 96: number analyzed (Participants) | 8 | 2
  Change at Week 96 | 0.0409 (0.03805) | 0.0607 (0.03585)
  Change at Week 120: number analyzed (Participants) | 8 | 3
  Change at Week 120 | 0.0173 (0.03303) | 0.0653 (0.02380)

15. Secondary Outcome: Number of Participants With Blood Transfusions or Thromboses
Description: Data was reported for number of participants for whom blood transfusion was required or who experienced the thrombosis events.
Time Frame: From first dose of study drug up to 3 weeks after last dose (Week 147)
Population: Participants in the mITT population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 12 | 7
Participants
  Blood transfusions | 3 | 4
  Thromboses | 0 | 0

16. Secondary Outcome: Number of Blood Transfusions
Description: Number of blood transfusions were reported.
Time Frame: From first dose of study drug up to 3 weeks after last dose (Week 147)
Population: Participants from mITT population who required blood transfusions.
Measure: Number; unit: Number of blood transfusions
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 3 | 4
Number of blood transfusions | 13 | 25

17. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale Total Score
Description: The FACIT-Fatigue scale questionnaire was used to determine the level of fatigue experienced by participants. This questionnaire was a 13-item measure that assessed self-reported fatigue and its impact upon daily activities and function. Item scores ranged from 0 ("not at all") to 4 ("very much"), and the total score ranged from 0 to 52, with higher scores indicating greater quality of life.
Time Frame: Baseline, Weeks 24, 48, 72, and 96
Population: Participants in the mITT population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | C5-INH Naïve Group | C5-INH Inadequate Response Group
Number analyzed (Participants) | 11 | 7
Scores on a scale
  Baseline | 43.82 (9.400) | 40.14 (13.533)
  Change at Week 24 | 0.09 (4.110) | -3.36 (8.066)
  Change at Week 48: number analyzed (Participants) | 8 | 3
  Change at Week 48 | -0.63 (2.387) | 2.33 (3.215)
  Change at Week 72: number analyzed (Participants) | 8 | 3
  Change at Week 72 | -0.38 (2.875) | -4.64 (12.016)
  Change at Week 96: number analyzed (Participants) | 8 | 3
  Change at Week 96 | -1.13 (4.357) | -18.00 (27.185)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 3 weeks after last dose (Week 147)
Description: The safety analysis population included all participants who received at least 1 capsule or tablet of study drug.
Groups:
- Complement Component 5 (C5) Inhibitor (C5-INH) Naïve Group: This group included participants who, prior to enrolling in their previous BCX9930 study, were either naïve to eculizumab or ravulizumab treatment, or naive to treatment with any complement inhibitor therapy (or had received no treatment in the prior 12 months), and with anemia due to ongoing intravascular hemolysis. Participants were to commence treatment at the same BCX9930 dose level and regimen last administered to that individual in the prior study. Per last protocol amendment, all participants received BCX9930 400 mg orally BID. Treatment duration was up to 144 weeks.
Arm/Group | Complement Component 5 (C5) Inhibitor (C5-INH) Naïve Group | C5-INH Inadequate Response Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 6/12 | 3/7
Other Adverse Events (participants affected / at risk) | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complement Component 5 (C5) Inhibitor (C5-INH) Naïve Group (N=12) | C5-INH Inadequate Response Group (N=7)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Boutonneuse fever (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complement Component 5 (C5) Inhibitor (C5-INH) Naïve Group (N=12) | C5-INH Inadequate Response Group (N=7)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (6)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 1 (2)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (7) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 2 (9)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 4 (5) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (10) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 5 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 3 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Creatinine urine increased (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 4 (12)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (8)
Influenza like illness (General disorders) | 1 (1) | 2 (3)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 2 (2)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (2)
Feeling abnormal (General disorders) | 0 (0) | 1 (3)
Oedema (General disorders) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (3)
Depression (Psychiatric disorders) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 1 (2) | 4 (5)
Chromaturia (Renal and urinary disorders) | 0 (0) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Maternal exposure via partner during pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (8)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (3)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The sponsor decided to prematurely terminate the study due to business reasons. Per change in planned analysis, data were analyzed and reported for safety and selected efficacy parameters (assessment of various clinical PNH symptoms severity, incidence of thromboembolic events, change from baseline in clinical measurements of PNH [LDH, hemoglobin, haptoglobin, reticulocytes, transfusion requirements], and change from baseline in FACIT]).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04702568/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04702568/SAP_001.pdf